CLINICAL TRIAL: NCT03378245
Title: Telemedicine-based, Multidisciplinary-team, Intervention to Reduce Unnecessary Hospitalizations and Healthcare Costs in Appalachia KY Skilled Nursing Facilities
Brief Title: Telemedicine-based, Multidisciplinary-team, Intervention to Reduce Unnecessary Hospitalizations
Acronym: TeleNH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Ronan Murphy (Other)
Responsible Party: Sponsor-Investigator, Richard Ronan Murphy, Assistant Professor of Neurology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: 13-0664-P3H
Record Dates: First submitted 2017-08-16; First posted 2017-12-19 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Dementia Alzheimers; Disruptive Behavior
MeSH Terms: conditions — Alzheimer Disease; Problem Behavior | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine Intervention (Experimental): Multidisciplinary telemedicine education of staff and providers on best practices for behavioral modification as well as education on best practices for pharmacologic therapies.
  Interventions: Behavioral: Behavioral modification and education on pharmacologic treatments.

INTERVENTIONS:
Behavioral: Behavioral modification and education on pharmacologic treatments. — Education and counseling of care-giving staff on behavioral modification strategies, as well as education about current standard of care best practices for pharmacologic interventions.

SUMMARY:
The purpose of this study is to investigate the use of telemedicine-based intervention at urban and rural skilled nursing facilities to recommend multidisciplinary dementia care to residents with dementia who are at risk for unnecessary hospitalization due behavioral or neuropsychiatric symptoms and/or complications as well as caregivers and facility staff. The multidisciplinary team is comprised of trained behavioral neurologists, social workers, advanced practice providers, primary medical team and nurse coordinators.

ELIGIBILITY:
Inclusion Criteria:

Dementia Care facility resident Problematic behavioral problems

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in the Neuropsychiatric Inventory (NPI) total score | 6 months
  The NPI assesses 10 behavioral symptom domains, scoring is based on symptom frequency and severity. The total NPI score sums the products of frequency and severity scores for each domain. Higher scores indicate more behavioral disturbance

SECONDARY OUTCOMES:
Change in the Resource Utilization in Dementia - Formal Care (RUD-FOCA) | 6 months
  The RUD-FOCA records the care time in three areas: activities of daily living (ADL), instrumental activities of daily living (IADL) and supervision.
Change in Quality of Life in Alzheimers Dementia (QoL-AD) | 6 months.
  13 quality of life items are rated on a four point scale, with 1 being poor and 4 being excellent. Total scores range from 13 to 52. It generally takes caregivers about 5 minutes to complete the measure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No